CLINICAL TRIAL: NCT06299956
Title: Supervised Exercise-based Rehabilitation for People With Intermittent Claudication - Study Protocol for a Danish Implementation Process (StRiDE).
Brief Title: Supervised Exercise-based Rehabilitation for People With Intermittent Claudication in Denmark
Acronym: StRiDE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Slagelse Hospital (Other)
Collaborators: Region Zealand (Other); Vordingborg Municipality (Unknown); Kalundborg municipality (Unknown); Køge Municipality (Unknown); Næstved municipality (Unknown); Solrød Municipality (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2023-SFHHB-IC-001
Record Dates: First submitted 2024-03-01; First posted 2024-03-08 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Intermittent Claudication
Keywords: Exercise therapy; Smoking cessation; Implementation; Stakeholders; Walking; Treadmill
MeSH Terms: conditions — Intermittent Claudication; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- The intervention group (Other): Supervised exercise therapy. Walking on a treadmill 3 times a week, for 12 weeks. Supervised by a physiotherapist.
  Interventions: Other: Supervised exercise therapy

INTERVENTIONS:
Other: Supervised exercise therapy — Walking on a treadmill at increasing elevation and pace.

SUMMARY:
The goal of this project is to implement a protocol for a supervised exercise therapy intervention including smoking cessation in the municipalities in region Zealand in Denmark. The participants are adults with intermittent claudication.

The objective of this project is to describe:

1. The development and design of the implementation process of a rehabilitative intervention including SET and smoking cessation in Region Zealand with a 6-month follow-up period after completion of the SET.
2. The ongoing quality monitoring process of the implementation in terms of referral, recruitment, retention, data completeness, intervention delivery and attendance and to collect feedback that will guide refinements of the intervention delivery and data collection.
3. Outcomes available for assessment of benefits and harms from the SET intervention.

Participants will be asked to do supervised exercise therapy by walking on a treadmill for 3 times a week for 12 weeks, and engage in smoking cessation, if they are smoking.

ELIGIBILITY:
Inclusion criteria:

* Relevant symptoms of intermittent claudication; leg pain when walking due to arteriosclerosis and relieve of symptoms during rest.
* Distal blood pressure with an ankle-brachial index (ABI) > 50 mmHg for non-diabetics or toe brachial index (TBI) > 40 mmHg for diabetics.

Exclusion criteria:

• Evaluated by a vascular surgeon: patients with contraindications e.g. medical issues or comorbidity that enables a participation in SET are not referred.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Maximal Walking Distance | Baseline, 12 weeks and 6 months from end of intervention
  Treadmill test 3.2 km/h and 0% inclination for 2 min. Then the inclination will incline 2% every 2 min until the patient cannot walk further. The distance is noted in meters.

SECONDARY OUTCOMES:
Pain-free walking distance | Baseline, 12 weeks and 6 months from end of intervention
  Treadmill test 3.2 km/h and 0% inclination for 2 min. Then the inclination will incline 2% every 2 min until onset of claudication pain(2-5 on claudication pain scale) The claudication scale is 1-5. First experienced claudication pain(2-5) is noted in meters.
Vascular Quality of Life Questionnaire-6 (VASCUQoL-6) | Baseline, 12 weeks and 6 months from end of intervention
  Patient reported questionnaire: Health-related quality of life. Each question is scored 1-4. When using the VQ6, the sum of each individual question score is used to generate a 'Total' Quality of Life Score (ranging from minimum 6 to maximum 24). A higher value indicates better health status.

CONTACTS AND LOCATIONS:
Overall Officials: Helle Bøgard, Principal Investigator — Slagelse Hospital
Locations (1):
- PROgrez, Slagelse, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hajdu SF, Bogard H, Aagaard TV, Roikjaer SG, Simony C, Dalhoff A, Houlind K, Luijk A, Ulriksen I, Jensen LT, Skou ST, Tang LH. Supervised exercise-based rehabilitation for people with intermittent claudication-Study protocol for a Danish implementation process (StRiDE). PLoS One. 2025 Jan 13;20(1):e0315577. doi: 10.1371/journal.pone.0315577. eCollection 2025. PMID 39804879